CLINICAL TRIAL: NCT03861273
Title: Phase 3, Open-label, Single-arm Study to Evaluate Efficacy and Safety of FIX Gene Transfer With PF-06838435 (rAAV-Spark100-hFIX-R338L) in Adult Male Participants With Moderately Severe to Severe Hemophilia B (FIX:C ≤2%) (BeneGene-2)
Brief Title: A Study to Evaluate the Efficacy and Safety of Factor IX Gene Therapy With PF-06838435 in Adult Males With Moderately Severe to Severe Hemophilia B
Acronym: BENEGENE-2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0371002; 2022-502844-11-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hemophilia B
Keywords: PF 06838435; Hemophilia; Hemophilia B; Factor IX; FIX; Gene Therapy; Infusion; rAAV Spark100 hFIX Padua; rAAV Spark100-hFIX-R338L; R338L; BeneGene 2; Hematological Diseases; Annualized bleeding rate (ABR)
MeSH Terms: conditions — Hemophilia B; Hemophilia A; Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PF-06838435/ fidanacogene elaparvovec (Experimental)
  Interventions: Biological: PF-06838435/ fidanacogene elaparvovec

INTERVENTIONS:
Biological: PF-06838435/ fidanacogene elaparvovec — Gene Therapy

SUMMARY:
This study will evaluate the efficacy and safety of PF-06838435 (a gene therapy drug) in adult male participants with moderately severe to severe hemophilia B (participants that have a Factor IX circulating activity of 2% or less). The gene therapy is designed to introduce genetic material into cells to compensate for missing or non-functioning Factor IX. Eligible study participants will have completed a minimum 6 months of routine Factor IX prophylaxis therapy during the lead in study (C0371004). Participants will be dosed once (intravenously) and will be evaluated over the course of 6 years. The main objective of the study will evaluate the annualized bleeding rate [ABR] for participants treated with gene therapy versus standard of care (SOC) therapy (FIX prophylaxis replacement regimen).

ELIGIBILITY:
Inclusion Criteria

* Males who completed 6 months of Factor IX prophylaxis therapy during the lead-in study (C0371004) prior to providing consent at the screening visit for this study.
* Documented moderately severe to severe hemophilia B (Factor IX activity < =2%)
* Previous experience with FIX therapy (=>50 documented exposure days to a FIX protein product)
* Suspension of prophylaxis therapy for hemophilia B after administration of the study drug
* Laboratory values (hemoglobin, platelets and creatinine) within study specified limits
* Agree to contraception until components of the drug are eliminated from their body
* Capable of giving signed informed consent

Exclusion Criteria

* Anti-AAVRh74var neutralizing antibodies (nAb) titer above the established threshold (ie, positive for nAb).
* History of inhibitor to Factor IX or inhibitor detected during screening. Clinical signs or symptoms of decreased response to Factor IX
* Hypersensitivity to Factor IX replacement product or IV immunoglobulin administration
* History of chronic infection or other chronic disease
* Any conditions associated with increased thromboembolic risk
* Concurrent clinically significant major disease or condition unsuitable for participation and/or may interfere with the interpretation of study results
* Laboratory values at screening visit that are abnormal or outside acceptable study limits
* Current unstable liver or biliary disease
* Currently on antiviral therapy for hepatitis B or C
* Planned surgical procedure requiring Factor IX surgical prophylactic factor treatment 15 months from screening visit
* Use of restricted therapies (e.g., blood products, acetylsalicylic acid [aspirin] or ibuprofen, other investigational therapy, and by-passing agents)
* Previously dosed in a gene therapy research trial at any time or in an interventional clinical study within 12 weeks of screening visit
* Active hepatitis B or C; hepatitis B surface antigen, hepatitis B virus deoxyribonucleic acid positivity, or hepatitis C virus ribonucleic acid positivity
* Significant liver disease
* Serological evidence of HIV1 or HIV2 infection with either CD4+ cell count <=200 mm3 and/or a viral load >20 copies/mL
* Study and sponsor staff involved in the conduct of the study and their families
* Unable to comply with study procedures
* Sensitivity to heparin or heparin induced thrombocytopenia
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 51 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2031-02-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (59):
- United States (12):
  - University of California, San Francisco - Clinical Research Center, San Francisco, California
  - University of California, San Francisco - Outpatient Hematology Clinic, San Francisco, California
  - Hemophilia and Thrombosis Center at the University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Indiana Hemophilia & Thrombosis Center, Inc., Indianapolis, Indiana
  - Indiana Hemophilia and Thrombosis Center, Inc, Indianapolis, Indiana
  - St. Vincent Hospital & Health Care Center, Inc., Indianapolis, Indiana
  - Madison Radiological Group, Madison, Mississippi
  - Mississippi Center for Advanced Medicine, Madison, Mississippi
  - Center for Human Phenomic Science CHPS, Philadelphia, Pennsylvania
  - Center for Human Phenomic Science, Philadelphia, Pennsylvania
  - Investigational Drug Service, Philadelphia, Pennsylvania
  - Penn Blood Disorder Center, Philadelphia, Pennsylvania
- Australia (5):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - Royal Brisbane and Women's Hospital, Herston
- Brazil (4):
  - Centro Estadual de Hemoterapia e Hematologia Marcos Daniel Santos - Hemoes, Vitória, Espírito Santo
  - Centro de Hematologia e Hemoterapia - Hemocentro de Campinas - UNICAMP, Campinas, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, São Paulo
  - Instituto Estadual de Hematologia Arthur de Siqueira Cavalcanti- HEMORIO, Rio de Janeiro
- Canada (3):
  - McMaster University Medical Centre - Hamilton Health Sciences, Hamilton, Ontario
  - Juravinski Hospital - Hamilton Health Sciences, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- France (2):
  - Hopital Cardiologique Louis Pradel - CRTH, Bron
  - Hopital Necker, Paris
- Germany (5):
  - Vivantes Klinikum Friedrichshain, Berlin
  - Vivantes Klinikum im Friedrichshain, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Universitätsklinikum Bonn, Anstalt des öffentlichen Rechts, Bonn
  - Universitätsklinikum Bonn, Bonn
- General Hospital of Athens "LAIKO", 2nd Regional Blood Transfusion Center, Athens, Greece
- Italy (2):
  - Azienda Ospedaliero Universitaria Careggi, Florence
  - Azienda Ospedaliera Universitaria Federico II, Naples
- Japan (4):
  - Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Nara Medical University Hospital, Kashihara, Nara
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - National Center for Child Health and Development, Setagaya-ku, Tokyo
- Saudi Arabia (2):
  - King Abdulaziz Medical City-Ministry of national guard, Riyadh, Kingdom of Saudi Arabia
  - King Faisal Specialist Hospital and Research Centre, Riyadh
- Kyung Hee University Hospital at Gangdong, Seoul, South Korea
- Spain (2):
  - Hospital Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitari Vall d´Hebrón, Barcelona
- Sweden (2):
  - Skåne University Hospital, Department of Hematology, Oncology and Radiation Physics, Malmo
  - ApoEx AB, Malmo
- Taiwan (6):
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Chung Shan Medical University, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Turkey (Türkiye) (4):
  - Acibadem Adana Hospital, Adana
  - Gaziantep University Sahinbey Training and Research Hospital, Gaziantep
  - Istanbul University Oncology Institute, Istanbul
  - Ege University Medical Faculty Hospital, Izmir
- United Kingdom (4):
  - Newcastle upon Tyne Hospitals NHS FT, Newcastle upon Tyne, TYNE & WEAR
  - Glasgow Royal Infirmary, Glasgow
  - Guy's and St. Thomas' NHS Foundation Trust, London
  - Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Wojciechowski J, Gaitonde P, Hughes JH, Ravva P. Population Modeling of Factor IX Activity Following Administration of Fidanacogene Elaparvovec Gene Therapy in Participants with Hemophilia B. Clin Pharmacokinet. 2025 Oct;64(10):1531-1548. doi: 10.1007/s40262-025-01535-y. Epub 2025 Aug 1. PMID 40750723
- [Derived] Cuker A, Kavakli K, Frenzel L, Wang JD, Astermark J, Cerqueira MH, Iorio A, Katsarou-Fasouli O, Klamroth R, Shapiro AD, Hermans C, Ishiguro A, Leavitt AD, Oldenburg JB, Ozelo MC, Teitel J, Biondo F, Fang A, Fuiman J, McKay J, Sun P, Rasko JEJ, Rupon J; BENEGENE-2 Trial Investigators. Gene Therapy with Fidanacogene Elaparvovec in Adults with Hemophilia B. N Engl J Med. 2024 Sep 26;391(12):1108-1118. doi: 10.1056/NEJMoa2302982. PMID 39321362
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C0371002

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately severe to severe hemophilia B, who completed a minimum 6 months of routine Factor IX prophylaxis therapy during the lead-in study C0371004 (NCT03587116), were enrolled in this study.
Pre-assignment Details: A total of 51 participants were screened in this study and 45 participants received a single dose of PF-06838435 (fidanacogene elaparvovec). Results presented are for primary outcome measures and only those secondary measures whose analysis was complete on a data cutoff date of 16 November 2022 (primary completion date [PCD]).
Groups:
- PF-06838435: Participants received PF-06838435 infusion on Day 1 at a dose of 5*10^11 vector genomes per kilogram (kg) of body weight. Short term follow-up: Participants were followed up for 52 weeks/Year 1 post infusion. Long term follow-up: Participants were followed up from Year 2 to 6.
Period: Screening Phase (3 Weeks)
Arm/Group | PF-06838435
Started | 51
Completed | 45
Not Completed | 6
Not completed — Other | 1
Not completed — Screen failure | 5
Period: Treatment Phase (Day 1)
Arm/Group | PF-06838435
Started | 45
Completed | 45
Not Completed | 0
Period: Follow-up Phase (Year 1)
Arm/Group | PF-06838435
Started | 45
Completed | 43
Not Completed | 2
Not completed — Ongoing | 2
Period: Long-Term Follow-Up (Year 2 to Year 6)
Arm/Group | PF-06838435
Started | 43
Completed | 0
Not Completed | 43
Not completed — Ongoing | 42
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants enrolled in the study and who received PF-06838435 infusion.
Groups:
- PF-06838435: All participants enrolled in the study and who received PF-06838435 infusion.
Arm/Group | PF-06838435
Number analyzed (Participants) | 45
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.18 (10.947)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Annualized Bleeding Rate (ABR) for Total Bleeds (Treated and Untreated) From Week 12 to Month 15
Description: ABR = number of total bleeding episodes on study during the given time period) *365.25/ (Date of last day - date of first day +1) in that time period. Surgical procedures were excluded from summary/analyses. Treated Bleed: An event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding (protocol definition, unless specifically referring to untreated bleed). Untreated Bleed: A bleeding event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002.
Time Frame: Pre-infusion period: minimum of 6 months through first dose of current study, an average of 1.31 years (FIX Prophylaxis arm); Week 12 to Month 15 post infusion in current study (PF-06838435 arm)
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (95% Confidence Interval); unit: Total bleeds per year
Groups:
- FIX Prophylaxis: Participants who received routine Factor IX (FIX) prophylaxis replacement therapy during the lead-in study C0371004. Participants subsequently received PF-06838435 infusion. This reporting arm served as control and it used data from lead-in study C0371004 for comparing data from the current study C0371002.
- PF-06838435: Eligible participants enrolled in the current study C0371002 and who received PF-06838435 infusion on Day 1. This reporting arm served as experimental arm.
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
Total bleeds per year | 4.43 [1.81 to 7.05] | 1.30 [0.59 to 2.02]
Statistical Analysis 1: Comparison: FIX Prophylaxis vs PF-06838435; Test type: Non-Inferiority — A repeated measure negative binomial regression model was used to do the hypothesis test on non-inferiority with one-sided test; p = 0.0081, Generalized linear model (GLM); The treatment difference and P-value were obtained from a repeated measures GLM with negative binomial distribution and identity link function; Mean Difference (Final Values) = -3.13, 95% CI 2-sided [-5.44 to -0.81]

2. Secondary Outcome: ABR for Treated Bleeds From Week 12 to Month 15
Description: ABR = number of total bleeding episodes on study during the given time period) *365.25/ (Date of last day - date of first day +1) in that time period. Surgical procedures were excluded from summary/analyses. Treated Bleed: An event necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding (protocol definition, unless specifically referring to untreated bleed). This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002.
Time Frame: as for outcome 1
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (95% Confidence Interval); unit: Treated bleeds per year
Groups:
- FIX Prophylaxis: Participants who received routine Factor IX (FIX) prophylaxis replacement therapy during the lead-in study (C0371004. Participants subsequently received PF-06838435 infusion. This reporting arm served as control and it used data from lead-in study C0371004 for comparing data from the current study C0371002.
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
Treated bleeds per year | 3.35 [1.71 to 4.98] | 0.73 [0.25 to 1.21]
Statistical Analysis 1: Comparison: FIX Prophylaxis vs PF-06838435; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; p = 0.0019, Generalized linear model (GLM); [statistical method as in outcome 1, analysis 1]; Median Difference (Final Values) = -2.62, 95% CI 2-sided [-4.27 to -0.96]

3. Secondary Outcome: Annualized Infusion Rate (AIR) of Exogenous FIX From Week 12 to Month 15
Description: AIR = number of exogenous infusions (for any reason) received during given time period *365.25/ (Date of last day - date of first day +1) in that time period. This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002.
Time Frame: as for outcome 1
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (Standard Deviation); unit: Exogenous infusions per year
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
Exogenous infusions per year | 58.83 (29.056) | 4.46 (10.028)
Statistical Analysis 1: Comparison: FIX Prophylaxis vs PF-06838435; The treatment difference (PF-06838435 - FIX Prophylaxis) estimate (95% CI) and p-value were obtained from paired t-test; Test type: Superiority; p < .0001, Paired t-test; Mean Difference (Final Values) = -54.37, 95% CI 2-sided [-63.64 to -45.10]

4. Secondary Outcome: Steady State Circulating Factor IX (FIX:C) From Week 12 to Month 15
Description: The certified central clinical laboratory analyzed the sample by two one-stage assays and a chromogenic assay. The first one-stage assay was performed on BCSXP analyzer with Actin-FSL reagent. The second one-stage assay used the same analyzer but SynthAsil as reagent. Data reported in this Outcome Measure is the geometric mean of all assessments from week 12 to Month 15.
Time Frame: Week 12 to Month 15
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion. The assessments at the visits following participant withdrawal/dropout/FIX prophylaxis resumption were imputed as 1.9%. Here, "Number Analyzed" signifies number of participants evaluable for specified rows of respective arms.
Measure: Geometric Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | PF-06838435
Number analyzed (Participants) | 45
Percentage of Normal
  Week 12 to Month 15: One-stage Assay (Actin-FSL Reagent) | 12.62 (8.92)
  Week 12 to Month 15: One-stage Assay (SynthASil Reagent) | 25.90 (16.89)
  Week 12 to Month 15: Chromogenic Assay | 13.49 (10.40)
Statistical Analysis 1: Comparison: PF-06838435; Week 12 to Month 15; Test type: Other; p < .0001, One-sided t-statistic testing — P-value from one-sided t-statistic testing the log transformation of the steady state FIX:C > log(5). Cumulative for 3 assays

5. Secondary Outcome: Circulating Factor IX (FIX:C) at Week 12, Week 24, Week 65
Description: The certified central clinical laboratory analyzed the sample by two one-stage assays and a chromogenic assay. The first one-stage assay was performed on BCSXP analyzer with Actin-FSL reagent. The second one-stage assay used the same analyzer but SynthAsil as reagent.
Time Frame: Week 12, Week 24, Week 65
Population: Dosed analysis set: participants enrolled in the study who received PF-06838435 infusion. The assessments at the visits following participant withdrawal/dropout/FIX prophylaxis resumption were imputed as 1.9%. "Number Analyzed": at each row represents the number of participants with valid FIX:C assessments at the respective time points. All participants reported under 'Number of Participants Analyzed' contributed data to the table; however, may not have evaluable data for every row.
Measure: Mean (Standard Deviation); unit: Percentage of Normal
Arm/Group | PF-06838435
Number analyzed (Participants) | 45
Percentage of Normal
  Week 12: One-stage Assay (Actin-FSL Reagent): number analyzed (Participants) | 43
  Week 12: One-stage Assay (Actin-FSL Reagent) | 13.52 (8.134)
  Week 12: One-stage Assay (SynthASil Reagent): number analyzed (Participants) | 44
  Week 12: One-stage Assay (SynthASil Reagent) | 27.79 (15.226)
  Week 12: Chromogenic Assay: number analyzed (Participants) | 44
  Week 12: Chromogenic Assay | 13.91 (9.302)
  Week 24: One-stage Assay (Actin-FSL Reagent): number analyzed (Participants) | 41
  Week 24: One-stage Assay (Actin-FSL Reagent) | 13.10 (11.144)
  Week 24: One-stage Assay (SynthASil Reagent): number analyzed (Participants) | 39
  Week 24: One-stage Assay (SynthASil Reagent) | 27.67 (21.340)
  Week 24: Chromogenic Assay: number analyzed (Participants) | 40
  Week 24: Chromogenic Assay | 14.83 (12.961)
  Week 65: One-stage Assay (Actin-FSL Reagent): number analyzed (Participants) | 34
  Week 65: One-stage Assay (Actin-FSL Reagent) | 13.10 (12.792)
  Week 65: One-stage Assay (SynthASil Reagent): number analyzed (Participants) | 35
  Week 65: One-stage Assay (SynthASil Reagent) | 27.47 (25.739)
  Week 65: Chromogenic Assay: number analyzed (Participants) | 35
  Week 65: Chromogenic Assay | 15.82 (16.996)

6. Secondary Outcome: Annualized Factor IX (FIX) Consumption From Week 12 to Month 15
Description: Annualized FIX consumption was reported by International Units per kilogram (IU/kg). This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002. Data reported in this Outcome Measure is average of all assessments from Week 12 to Month 15.
Time Frame: as for outcome 1
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (Standard Deviation); unit: IU/kg per year
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
IU/kg per year | 3170.74 (1634.753) | 235.04 (538.977)
Statistical Analysis 1: Comparison: FIX Prophylaxis vs PF-06838435; Test type: Superiority; p < .0001, Paired t-test; Mean Difference (Final Values) = -2935.70, 95% CI 2-sided [-3403.10 to -2468.30]

7. Secondary Outcome: ABR for Spontaneous Bleeds From Week 12 to Month 15
Description: ABR = number of total bleeding episodes on study during the given time period) *365.25/ (Date of last day - date of first day +1) in that time period. Surgical procedures were excluded from summary/analyses. Surgical procedures were excluded from summary/analyses. Spontaneous Bleeds: Bleeding for no apparent/known reason particularly into the joints, muscles, and soft tissues. This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002.
Time Frame: as for outcome 1
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (95% Confidence Interval); unit: Spontaneous bleeds per year
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
Spontaneous bleeds per year | 3.24 [0.92 to 5.56] | 0.69 [0.19 to 1.20]
Statistical Analysis 1: Comparison: FIX Prophylaxis vs PF-06838435; Test type: Non-Inferiority — The treatment difference and P-value were obtained from a repeated measures GLM with negative binomial distribution and identity link function; p = 0.0191, Generalized linear model (GLM); Mean Difference (Final Values) = -2.55, 95% CI 2-sided [-4.67 to -0.42]

8. Secondary Outcome: ABR for Traumatic Bleeds From Week 12 to Month 15
Description: ABR = number of total bleeding episodes on study during the given time period) *365.25/ (Date of last day - date of first day +1) in that time period. Surgical procedures were excluded from summary/analyses. Surgical procedures were excluded from summary/analyses. Traumatic Bleeds: Bleeding event occurring for an apparent/known reason. This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002.
Time Frame: as for outcome 1
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (95% Confidence Interval); unit: Traumatic bleeds per year
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
Traumatic bleeds per year | 1.16 [0.34 to 1.98] | 0.59 [0.26 to 0.92]
Statistical Analysis 1: Comparison: FIX Prophylaxis vs PF-06838435; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p = 0.1528, Generalized linear model (GLM); Median Difference (Final Values) = -0.57, 95% CI 2-sided [-1.35 to 0.21]

9. Secondary Outcome: ABR for Untreated Bleeds From Week 12 to Month 15
Description: ABR = number of total bleeding episodes on study during the given time period) *365.25/ (Date of last day - date of first day +1) in that time period. Surgical procedures were excluded from summary/analyses. Surgical procedures were excluded from summary/analyses. Untreated Bleed: A bleeding event not necessitating administration of coagulation factor within 72 hours of signs or symptoms of bleeding. This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002.
Time Frame: as for outcome 1
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (95% Confidence Interval); unit: Untreated bleeds per year
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
Untreated bleeds per year | 1.07 [-0.32 to 2.47] | 0.57 [0.14 to 1.00]
Statistical Analysis 1: Comparison: FIX Prophylaxis vs PF-06838435; Test type: Non-Inferiority — [test comment as in outcome 7, analysis 1]; p = 0.3738, Generalized linear model (GLM); Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-1.63 to 0.61]

10. Secondary Outcome: Number of Target Joint Bleeds From Week 12 to Month 15
Description: Target Joint: Defined as a major joint (e.g., hip, elbow, wrist, shoulder, knee, and ankle) into which repeated bleeds occurred (three or more spontaneous bleeds into a single joint within a consecutive 6-month period). A target joint was considered resolved when there were =<2 bleeds into the joint within a 12-month period. Joint Bleed: A bleeding episode characterized by rapid loss of range of motion as compared with baseline that was associated with any combination of the following: pain or an unusual sensation in the joint, palpable swelling, and warmth of the skin over the joint. This outcome measure compared data collected from lead-in study C0371004 and from current study C0371002. Pre-infusion period = at least 6 months of prospectively collected data while receiving FIX prophylaxis replacement therapy in lead-in study C0371004 up to dosing in current study C0371002.
Time Frame: as for outcome 1
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Mean (Standard Deviation); unit: Target joint bleeds
Arm/Group | FIX Prophylaxis | PF-06838435
Number analyzed (Participants) | 45 | 45
Target joint bleeds | 2.9 (7.81) | 0.3 (1.02)

11. Secondary Outcome: Percentage of the Participants Without Bleeds From Week 12 to Month 15
Description: Percentage of participants without bleeds (total bleeds and treated bleeds) were summarized by type from Week 12 to Month 15.
Time Frame: Week 12 to Month 15
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion.
Measure: Number; unit: Percentage of participants
Arm/Group | PF-06838435
Number analyzed (Participants) | 45
Percentage of participants
  Without treated bleeds | 73.3
  Without treated and untreated bleeds | 64.4

12. Secondary Outcome: Change From Baseline in Joint Health as Measured by the Hemophilia Joint Health Score (HJHS) Instrument at Month 12
Description: A qualified healthcare professional assessed six joints (left ankle, right ankle, left elbow, right elbow, left knee, right knee) scored from 0 to 20 based on: duration of swelling, muscle atrophy, crepitus, flexion loss, extension loss, instability, joint pain, and strength. Gait was scored (0 to 4) based on walking, stairs, running, hopping on one leg. Total score = sum of scores from all joints + gait score ranged from 0 to 124, with the higher the number equating to more severe joint damage.
Time Frame: Baseline, Month 12
Population: Dosed analysis set included all participants enrolled in the study who received PF-06838435 infusion. Here, "Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows of respective arms.
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06838435
Number analyzed (Participants) | 44
Units on a scale
  Baseline | 17.8 [13.1 to 22.5]
  Change at Month 12: number analyzed (Participants) | 36
  Change at Month 12 | -2.6 [-4.7 to -0.6]
Statistical Analysis 1: Comparison: PF-06838435; Test type: Other; p = 0.0117, Paired t-test

13. Secondary Outcome: Change From Baseline in Hemophilia Quality of Life (Haem A QoL) Physical Health Domain at Month 12
Description: The Haem-A-QoL questionnaire contained 46 items with ten domains that assessed health in the following areas: Physical Health; Feelings; View of Self; Sports and Leisure; Work and School; Dealing with Haemophilia; Treatment; Future; Family Planning; and Partnership and Sexuality. The physical health domain was considered as the primary domain in this questionnaire, had a transformed score range from 0 to 100, with lower scores representing higher quality of life. In this Outcome Measure Physical Health domain scores of Haem A QoL are reported.
Time Frame: Baseline, Month 12
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06838435
Number analyzed (Participants) | 40
Units on a scale
  Baseline | 31.00 [23.02 to 38.98]
  Change at Month 12: number analyzed (Participants) | 37
  Change at Month 12 | -7.70 [-12.95 to -2.45]
Statistical Analysis 1: Comparison: PF-06838435; Test type: Other; p = 0.0052, Paired t-test

14. Secondary Outcome: Change From Baseline in Hemophilia Activities List (HAL) Complex Lower Extremity Activities Component Score at Month 12
Description: The HAL was a multiple domain measure of the impact of hemophilia on functional abilities in adults. The 7 domains of this instrument contained 42 items in total, as follows: lying/sitting/kneeling/standing; lower (leg) functioning; upper (arm) functioning; transportation; self-care; household tasks; and sports/leisure. Selected items from five of the domains were used to create three components: upper extremity; basic lower extremity; and complex lower extremity activities. The component score of "complex lower extremity activities" was the most important in this questionnaire, had a transformed score range from 0 to 100, higher values indicated less functional limitations in performing tasks.
Time Frame: Baseline, Month 12
Population: as for outcome 12
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | PF-06838435
Number analyzed (Participants) | 40
Units on a scale
  Baseline | 67.06 [59.10 to 75.02]
  Change at Month 12: number analyzed (Participants) | 37
  Change at Month 12 | 7.59 [1.07 to 14.11]
Statistical Analysis 1: Comparison: PF-06838435; Test type: Other; p = 0.0237, Paired t-test

15. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious TEAEs
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

16. Secondary Outcome: Number of Participants With Adverse Events of Special Interest
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

17. Secondary Outcome: Number of Participants With Positive Neutralizing Antibody (nAb) to Adeno-associated Virus Vector (AAV) and Anti-Drug Antibody (ADA)
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

18. Secondary Outcome: ABR for Total Bleeds (Treated and Untreated) Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

19. Secondary Outcome: ABR for Treated Bleeds Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

20. Secondary Outcome: AIR of Exogenous Factor IX Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

21. Secondary Outcome: FIX: C Level Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

22. Secondary Outcome: Annualized Factor IX Consumption Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

23. Secondary Outcome: ABR for Spontaneous and Traumatic, and Untreated Bleeds Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

24. Secondary Outcome: Change From Baseline in Joint Health as Measured by the HJHS Instrument Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Baseline, 6 years
Reporting Status: Not Posted, anticipated posting 2031-03

25. Secondary Outcome: Number of Target Joint Bleeds Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

26. Secondary Outcome: Change From Baseline in Haem A QoL Physical Health Domain Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Baseline, Maximum up to 6 years (Week 312) after PF-06838435 infusion
Reporting Status: Not Posted, anticipated posting 2031-03

27. Secondary Outcome: Change From Baseline in HAL Complex Lower Extremity Activities Component Score Through the Study
Description: Results would be posted at secondary completion date.
Time Frame: Baseline, 6 years
Reporting Status: Not Posted, anticipated posting 2030-03

ADVERSE EVENTS:
Time Frame: Day 1 up to analysis data cut-off 16-Nov-2022 (approximately 3 years 3 months)
Description: Same event may appear as both non-SAE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. All participants enrolled in the study and who received PF-06838435 infusion.
Groups:
- PF-06838435: All participants enrolled in the study and who received PF-06838435 infusion and have no significant interruption of efficacy measurement
Arm/Group | PF-06838435
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 7/45
Other Adverse Events (participants affected / at risk) | 37/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06838435 (N=45)
Anaemia (Blood and lymphatic system disorders) | 2
Duodenal ulcer (Gastrointestinal disorders) | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1
COVID-19 (Infections and infestations) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Pilonidal disease (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Coagulation factor IX level decreased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06838435 (N=45)
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 3
Hepatic function abnormal (Hepatobiliary disorders) | 6
Hepatic steatosis (Hepatobiliary disorders) | 3
COVID-19 (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 8
Upper respiratory tract infection (Infections and infestations) | 4
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 3
Hepatic enzyme increased (Investigations) | 3
SARS-CoV-2 test positive (Investigations) | 3
Transaminases increased (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 3
Acne (Skin and subcutaneous tissue disorders) | 3
Hypertension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
C0371004 lead-in ongoing study: did not involve any investigational intervention; designed to collect bleed, infusion data while participants were on their prophylaxis FIX therapy for a minimum of 6 months; data served as within participant comparison group for C0371002; participant flow and AEs are missing as the study has not concluded yet (some participants in the C0371004 are ongoing and supporting a different study NCT04370054) and data will be provided at conclusion of the lead-in study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/73/NCT03861273/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03861273/SAP_001.pdf